CLINICAL TRIAL: NCT04690192
Title: CNCT19 Following Autologous Stem Cell Transplantation in Patients With Relapsed or Refractory Aggressive B-cell Lymphoma
Brief Title: CNCT19 Following ASCT in Patients With Relapsed or Refractory B-cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020013
Record Dates: First submitted 2020-12-26; First posted 2020-12-30 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Large B-cell Lymphoma
Keywords: autologous stem-cell transplantation; anti-CD19 CAR T-cell; large B-cell lymphoma
MeSH Terms: interventions — Gemcitabine; Busulfan; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CNCT19 following ASCT (Experimental): Participants will receive high-dose chemotherapy followed by stem-cell reinfusion, and a fixed dose of CNCT19 (2×10^6/kg) will be infused in a single-dose on day +2, +3 or +4.
  Interventions: Biological: CNCT19; Drug: Gemcitabine Injection; Drug: busulfan; Drug: Melphalan Injection

INTERVENTIONS:
Biological: CNCT19 — 2×10^6/kg, infused in a single-dose on day +2, +3 or +4 following stem-cell infusion
Drug: Gemcitabine Injection — 600mg/m2/h, infused for 3 hours with loading bolus of 75mg/m2, day -7, -3,
Drug: busulfan — 105mg/m2, day -7 until -5,
Drug: Melphalan Injection — 60mg/m2, day -3, -2

SUMMARY:
The primary objective of this study is to explore the safety and efficacy of CNCT19 (a second-generation anti-CD19 CAR T-cell using 4-1BB as co-stimulatory domain provided by Juventas, Tianjin, China) infusion following ASCT in patients with relapsed or refractory B-cell lymphoma.

DETAILED DESCRIPTION:
This is a single-center, non-randomized, open-label, prospective clinical trial to evaluate the safety and efficacy of CNCT19 infusion following high-dose chemotherapy and autologous stem-cell transplantation (HDT/ASCT) in patients with relapsed or refractory B-cell lymphoma. CNCT19 cells will be infused on day +3 (±1d) with a fixed dose of 2×10^6/kg. The study will assess the safety and efficacy of this combinational therapy, including the incidence and severity of cytokine release syndrome (CRS), immune effector cell-associated neurotoxicity syndrome (ICANS), hematological, and other non-hematological toxicities, and objective response rates and complete response rates and survivals of the subjects.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed large B-cell lymphoma including the following types

   * diffuse large B-cell lymphoma
   * high-grade B-cell lymphoma with or without MYC and BLC2 and/or BCL6 rearrangement
   * transformed lymphoma
2. Relapsed or refractory diseases fulfilling one of the following criteria (individuals must have received anti-CD20 monoclonal antibody and anthracycline-containing chemotherapy regimen)

   * Primary refractory disease, defined as disease progression after first-line immunochemotherapy or disease progression within 6 weeks of the end of the last chemotherapy
   * Stable disease (SD) as best response after at least 4 cycles of first-line therapy
   * Partial response (PR) as best response after at least 6 cycles of first-line therapy (biopsy-proven residual disease is needed for individuals with Deauville score of 4)
   * PR as best response after at least 2 cycles of second-line therapy
   * Disease relapse ≤12 months after the completion of first-line immunochemotherapy
   * Relapsed or refractory disease after ≥2 lines of chemotherapy
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Adequate bone marrow function as evidenced by:

   * Absolute neutrophil count (ANC) ≥ 1000/uL
   * Platelet count≥ 75,000/uL
5. Adequate renal and hepatic function defined as:

   * Serum alanine aminotransferase (ALT/AST) ≤ 3 upper limit of normal (ULN)
   * Total bilirubin ≤1.5 mg/dL, except in individuals with Gilbert's syndrome
   * Serum creatinine ≤2 ULN, or creatinine clearance (as estimated by Cockcroft Gault) ≥ 40 mL/min
6. Cardiac ejection fraction ≥ 50%
7. Baseline oxygen saturation > 92% on room air
8. Life expectancy ≥3 months

Key Exclusion Criteria:

1. Active Central Nervous System (CNS) involvement by lymphoma
2. History of autologous or allogeneic stem cell transplantation
3. Active HBV or HCV infection, defined as HBV-DNA or HCV-DNA levels above the normal upper limit, with or without abnormal liver function. Individuals with positive HBsAg or HBcAb should receive antiviral prophylaxis for at least 12 months after CNCT19 infusion.
4. Presence of uncontrolled infection, cardio-cerebrovascular disease，coagulopathy, or connective tissue disease.
5. History of seizure or other CNS disorder
6. History of HIV infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Percentage of participants experiencing adverse events | from the first day of high-dose chemotherapy until 2 years post CNCT19 infusion

SECONDARY OUTCOMES:
Complete Response (CR) Rate | 2 years post CNCT19 infusion
  Complete Response rate is defined as the incidence of a CR per the Lugano Classification (Cheson et al, 2014), as determined by study investigators.
Objective Response Rate (ORR) | 2 years post CNCT19 infusion
  ORR is defined as the incidence of either a CR or a partial response (PR) per the Lugano Classification as determined by study investigators.
Progression-Free Survival (PFS) | 2 years post CNCT19 infusion
  PFS is defined as the time from the CNCT19 infusion date to the date of disease progression or death from any cause.
Duration of Response (DOR) | 2 years post CNCT19 infusion
  DOR is defined only for participants who experience an objective response after CNCT19 infusion and is the time from the first objective response to disease progression or death from any cause.
Disease-Free Survival (DFS) | 2 years post CNCT19 infusion
  DFS is defined only for participants who achieve complete response after CNCT19 infusion and is the time from complete response to disease progression or death from any cause.
Overall Survival (OS) | 2 years post CNCT19 infusion
  OS is defined as the time from CNCT19 infusion to the date of death from any cause.

OTHER OUTCOMES:
Levels of CNCT19 in blood | 2 years post CNCT19 infusion
Levels of cytokines in serum | 1 month post CNCT19 infusion
Levels of lymphocyte subsets in blood | 1 year post CNCT19 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Dehui Zou, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, CAMS & PUMC
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: The data from this study can be accessed for up to two years, starting two years after the completion of the research.
Access Criteria: The IPD are available from the principle investigator on reasonable request.

REFERENCES:
- [Derived] Liu W, Liu W, Zou H, Chen L, Huang W, Lv R, Xu Y, Liu H, Shi Y, Wang K, Wang Y, Xiong W, Deng S, Yi S, Sui W, Peng G, Ma Y, Wang H, Lv L, Wang J, Wei J, Qiu L, Zheng W, Zou D. Combinational therapy of CAR T-cell and HDT/ASCT demonstrates impressive clinical efficacy and improved CAR T-cell behavior in relapsed/refractory large B-cell lymphoma. J Immunother Cancer. 2024 Apr 16;12(4):e008857. doi: 10.1136/jitc-2024-008857. PMID 38631712